CLINICAL TRIAL: NCT07171931
Title: Comparison of the Postoperative Analgesic Efficacy of Genicular Block and IPACK Block in Addition to Adductor Canal Block in Knee Arthroplasty
Brief Title: Genicular vs IPACK Block for Analgesia in Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAD-FR-42
Record Dates: First submitted 2025-08-27; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management in Total Knee Arthroplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPACK Group (Active Comparator): Patients who will receive IPACK block
  Interventions: Procedure: IPACK block
- Genicular Group (Active Comparator): Patients who will receive genicular block
  Interventions: Procedure: Genicular nerve block with bupivacaine

INTERVENTIONS:
Procedure: IPACK block — After the general anesthesia induction, IPACK block will be performed with 0.25% bupivacaine (20 mL) using ultrasound in addition to adductor canal block.
  Arms: IPACK Group
Procedure: Genicular nerve block with bupivacaine — After the general anesthesia induction, genicular block will be performed with 0.25% bupivacaine (20 mL) using ultrasound in addition to adductor canal block.
  Arms: Genicular Group

SUMMARY:
Total knee arthroplasty (TKA) is one of the most frequently performed orthopedic procedures, and with the aging population, the global number of TKA cases is expected to increase sixfold within the next decade. Postoperative pain following TKA is often severe and difficult to manage, which may increase the risk of developing chronic pain. Effective pain control is therefore a major concern, and multimodal analgesia is recommended to enhance analgesia, reduce opioid consumption, and minimize opioid-related side effects.

Peripheral nerve blocks (PNBs) are an integral part of multimodal regimens. Among them, the adductor canal block (ACB), which provides analgesia to the anteromedial aspect of the knee while preserving motor function, is widely used. The optimal analgesic strategy for TKA should not only ensure adequate pain relief but also maintain quadriceps strength to allow early mobilization. Motor-sparing blocks combined with multimodal analgesia have become increasingly popular because they facilitate early rehabilitation, decrease opioid requirements, and improve recovery outcomes.

The knee joint has a complex innervation, receiving contributions from the femoral, sciatic, and obturator nerves. For this reason, combining different PNBs may provide superior analgesia compared to a single block (2). The genicular nerves, consisting of branches from the femoral, common peroneal, saphenous, tibial, and obturator nerves, innervate the knee capsule. Genicular nerve block specifically targets these branches and has been used to manage postoperative pain in TKA patients.

Another motor-sparing option is the interspace between the popliteal artery and posterior capsule of the knee (IPACK) block, which provides analgesia to the posterior aspect of the knee. Using ultrasound guidance, local anesthetic is deposited between the posterior capsule and the popliteal artery. This approach spares the main trunks of the tibial and common peroneal nerves while effectively blocking the terminal branches innervating the posterior capsule, including the genicular nerves and the popliteal plexus.

However, there are no studies in the literature directly comparing IPACK and genicular blocks. With this study, the investigators aim to compare the efficacy of these two blocks in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total knee arthroplasty
* ASA physical status I-III

Exclusion Criteria:

* BMI > 35
* Patients < 50 kg
* Allergy to study medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative day 1 (24th hour)
  Amount of morphine in the postoperative period (mg)

SECONDARY OUTCOMES:
NRS Scores | Postoperative day 1 (1st, 6th, 12th and 24th hour)
  Numeric Rating Scale scores, between 0-10 (0= no pain, 10=worst pain imaginable)
QoR-15 | Postoperative 12th day
  Quality of Recovery-15: 15-item questionnaire that assesses patients' overall quality of recovery, between 0-150.
Nausea-vomiting | Postoperative day 1
  Number of patients who has nausea or vomiting
Rescue analgesic | Postoperative day 1
  The use of rescue analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Ufuk Yörükoğlu, Principal Investigator — Kocaeli University

IPD SHARING:
Plan to Share IPD: No